CLINICAL TRIAL: NCT04366622
Title: Investigation of Pharmacokinetics, Safety, and Tolerability of BAY 63-2521 in Male and Female Subjects With Hepatic Impairment (Classified as Child Pugh A or B) and in Age-, Weight- and Gender-matched Healthy Subjects Following a Single Oral Dose of 1 mg BAY 63-2521 in a Single-center, Non-randomized, Non-controlled, Non-blinded, Observational Study With Group Stratification
Brief Title: Study on the Safety of BAY 63-2521, How it is Tolerated and the Way the Body Absorbs, Distributes and Gets Rid of the Study Drug Given as a Single Oral Dose of 1 mg Tablet in Participants With Impaired Liver Function and Healthy Participants Matched for Age-, Gender-, and Weight
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 15001; 2009-017684-42 (EudraCT Number)
Record Dates: First submitted 2020-04-23; First posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Clinical Pharmacology
MeSH Terms: interventions — riociguat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Riociguat, Child Pugh A (Experimental): Participants with liver cirrhosis and mild hepatic impairment received a single dose of 1 mg (2 x 0.5 mg IR tablet) of riociguat in the fasted state
  Interventions: Drug: Riociguat (Adempas, BAY 63-2521)
- Riociguat, Child Pugh B (Experimental): Participants with liver cirrhosis and moderate hepatic impairment received a single dose of 1 mg (2 x 0.5 mg IR tablet) of riociguat in the fasted state
  Interventions: Drug: Riociguat (Adempas, BAY 63-2521)
- Riociguat, control A (Experimental): Healthy age-, weight-, and gender- matched participants to Child Pugh A group received a single dose of 1 mg (2 x 0.5 mg IR tablet) of riociguat in the fasted state
  Interventions: Drug: Riociguat (Adempas, BAY 63-2521)
- Riociguat, control B (Experimental): Healthy age-, weight-, and gender- matched participants to Child Pugh B group received a single dose of 1 mg (2 x 0.5 mg IR tablet) of riociguat in the fasted state
  Interventions: Drug: Riociguat (Adempas, BAY 63-2521)

INTERVENTIONS:
Drug: Riociguat (Adempas, BAY 63-2521) — 0.5 mg riociguat as an immediate-release (IR) tablet

SUMMARY:
BAY 63-2521 is intended to be used for a disease that affects the blood flow through the lungs. Renal impairment is a common condition in patients with this disease. The goal of the study is to learn more about the safety of BAY 63-2521, how it is tolerated and the way the body absorbs, distributes and gets rid of the study dug given as a single oral dose of 1 mg tablet in participants with renal impairment and healthy participants matched for age-, gender-, and weight

ELIGIBILITY:
Inclusion criteria for all subjects:

* Male and female White subjects 18 to ≤79 years of age, BMI between 18 and 34 kg/m^2
* Women without childbearing potential or with childbearing potential but only if the pregnancy test is negative and are under highly effective contraception

Inclusion criteria for subjects with liver cirrhosis:

* Documented liver cirrhosis confirmed by histopathology, eg previous liver biopsy, laparoscopy, or ultrasound Hepatic impairment (Child Pugh A or B)
* Stable liver disease

Inclusion criteria for healthy subjects:

- Age- (+/-10 years), weight- (+/-10 kg body weight), and gender-matched to a subject with liver cirrhosis as far as possible

Exclusion criteria for all subjects:

* Febrile illness within 1 week before the start of the study
* Hypersensitivity to riociguat and / or to inactive constituents
* Smoking

Exclusion criteria for subjects with liver cirrhosis:

* Hemoglobin <8 g/dL
* Severe cerebrovascular or cardiac disorders, eg myocardial infarction less than 6 months prior to dosing, congestive heart failure of NYHA grade III or IV, severe arrhythmia requiring antiarrhythmic treatment
* Evidence of hepatic encephalopathy related to chronic liver disease > Grade II
* Renal failure with a creatinine clearance <40 mL/min
* Resting heart rate in the awake subject below 45 BPM or above 100 BPM
* Systolic blood pressure (SBP) below 100 mmHg or above 160 mmHg, Diastolic blood pressure (DBP) above 95 mmHg
* Platelet count <30 x 10^9/L
* History of bleeding within the past 3 months
* AP >4 times the upper limit of normal (ULN)
* AST or ALT in conjunction with GGT >= 4 times the ULN (an isolated elevation of GGT >4 times ULN did not exclude the subject)
* Serum albumin <20 g/L
* Diabetes mellitus with a fasting blood glucose >220 mg/dL or HbA1c >10%
* Prothrombin time (Quick test) <30%
* Subjects who had undergone porto-caval shunt surgery
* Use of medications known to interfere with hepatic metabolism (eg cimetidine, barbiturates, phenothiazines, etc) or known to alter other major organs or systems within 30 days prior to dosing
* Severe infection, malignancy, psychosis, or any clinically significant illness within 4 weeks prior to dosing
* Concomitant use of any medication except medications necessary for the treatment of the kidney disease or related complications
* Concomitant use of phosphodiesterase-5 inhibitors, endothelin receptor antagonists (ERAs, eg bosentan), intravenous or inhalative prostacyclins, or nitrates
* Concomitant use of potent CYP3A4 and P-gp inhibitors

Exclusion criteria for healthy subjects:

* Conspicuous findings in medical history or pre-study examination
* History of relevant diseases of vital organs, central nervous system, or other organs
* Resting heart rate in the awake subject below 45 BPM or above 90 BPM
* SBP below 100 mmHg or above 145 mmHg, DBP above 95 mmHg
* Regular daily consumption of more than 1 liter of usual beer or the equivalent quantity of approximately 40 g of alcohol in another form

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-04-14; Primary Completion 2011-04-28 (Actual); Study Completion 2011-09-15 (Actual)

PRIMARY OUTCOMES:
AUC | Pre-dose and up to 72 hours post-dose, additionally up to 96 hours post-dose for Child Pugh B group only
  Area under the plasma concentration vs time curve from zero to infinity for total (bound and unbound) drug after single dose for BAY 63-2521 and its metabolite M1 (BAY 60-4552)
Cmax | Pre-dose and up to 72 hours post-dose, additionally up to 96 hours post-dose for Child Pugh B group only
  Maximum total (bound and unbound) drug concentration in plasma after single dose administration for BAY 63-2521 and its metabolite M1
t½ | Pre-dose and up to 72 hours post-dose, additionally up to 96 hours post-dose for Child Pugh B group only
  Half-life associated with the terminal slope for BAY 63-2521 and its metabolite M1
fu | From 2 hours post-dose up to 24 hours post-dose
  Fraction unbound for BAY 63-2521 and its metabolite M1
AUCu | From 2 hours post-dose up to 24 hours post-dose
  AUC for unbound drug for BAY 63-2521 and its metabolite M1
Cmax,u | From 2 hours post-dose up to 24 hours post-dose
  Cmax for unbound drug for BAY 63-2521 and its metabolite M1

SECONDARY OUTCOMES:
AUC/D | Pre-dose and up to 72 hours post-dose, additionally up to 96 hours post-dose for Child Pugh B group only
  AUC divided by dose (mg) for BAY 63-2521 and its metabolite M1
AUCnorm | Pre-dose and up to 72 hours post-dose, additionally up to 96 hours post-dose for Child Pugh B group only
  AUC divided by dose (mg) per kg body weight for BAY 63-2521 and its metabolite M1
AUCu,norm | From 2 hours post-dose up to 24 hours post-dose
  AUCnorm for unbound drug for BAY 63-2521 and its metabolite M1
AUC(0-tlast) | Pre-dose and up to 72 hours post-dose, additionally up to 96 hours post-dose for Child Pugh B group only
  AUC from time 0 to the last data point for BAY 63-2521 and its metabolite M1
Cmax/D | Pre-dose and up to 72 hours post-dose, additionally up to 96 hours post-dose for Child Pugh B group only
  Cmax divided by dose (mg) for BAY 63-2521 and its metabolite M1
Cmax,norm | Pre-dose and up to 72 hours post-dose, additionally up to 96 hours post-dose for Child Pugh B group only
  Cmax divided by dose (mg) per kg body weight for BAY 63-2521 and its metabolite M1
Cmax,u,norm | From 2 hours post-dose up to 24 hours post-dose
  Cmax,norm for unbound drug for BAY 63-2521 and its metabolite M1
tmax | Pre-dose and up to 72 hours post-dose, additionally up to 96 hours post-dose for Child Pugh B group only
  Time to reach maximum drug concentration in plasma after single dose for BAY 63-2521 and its metabolite M1
MRT | Pre-dose and up to 72 hours post-dose, additionally up to 96 hours post-dose for Child Pugh B group only
  Mean residence time for BAY 63-2521 and its metabolite M1
CL/F | Pre-dose and up to 72 hours post-dose, additionally up to 96 hours post-dose for Child Pugh B group only
  Total body clearance of total (bound and unbound) drug from plasma calculated after oral administration (apparent oral clearance) for BAY 63-2521 and its metabolite M1
CLu/F | From 2 hours post-dose up to 24 hours post-dose
  CL/F for unbound drug for BAY 63-2521 and its metabolite M1
Vz/F | Pre-dose and up to 72 hours post-dose, additionally up to 96 hours post-dose for Child Pugh B group only
  Apparent volume of distribution during terminal phase after oral administration for BAY 63-2521 and its metabolite M1
AE,ur | Pre-dose and up to 72 hours post-dose
  Amount of (total) drug excreted in urine for BAY 63-2521 and its metabolite M1
CLR | Pre-dose and up to 72 hours post-dose
  Renal body clearance of drug for BAY 63-2521 and its metabolite M1
Number of participants with adverse events | Approximately 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/